CLINICAL TRIAL: NCT06212271
Title: A Randomized, Placebo-Controlled Mechanistic Clinical Trial of Colchicine in Patients With Peripheral Artery Disease
Brief Title: Mechanistic Clinical Trial of Colchicine in Patients With Peripheral Artery Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 854429
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Artery Disease
Keywords: colchicine; atherosclerotic cardiovascular disease; peripheral artery disease; atherosclerosis; inflammation
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine (0.6 mg oral daily for 4-weeks) will be the drug administered in this study.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): This arm is a matching placebo that will be administered in the same fashion as the experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — See arm description.
  Arms: Colchicine
Drug: Placebo — See arm description.
  Arms: Placebo

SUMMARY:
The goal of this mechanistic clinical trial is to test the effects of reducing inflammatory signaling in femoral artery atherosclerotic plaques. Researchers will compare patients receiving colchicine to patients receiving placebo to determine the effect of colchicine on the inflammatory state of atherosclerotic femoral arteries.

DETAILED DESCRIPTION:
Patients with peripheral artery disease who will be undergoing femoral endarterectomy will be randomized 1:1 to receive colchicine (0.6mg oral) or placebo daily for 4 weeks prior to 18F-FDG PET/CT imaging. At the baseline visit, study procedures will be reviewed with eligible participants and the study team will obtain written informed consent. Baseline blood samples for laboratory studies will be collected and assayed, as well as additional blood samples for research. Participants will completed study questionnaires at baseline and at the imaging visit. Participants will receive follow-up phone calls with the study team. All eligible participants will be approached for participation in an imaging visit. At the imaging visit, participants will repeat laboratory tests and undergo non-invasive molecular imaging to evaluate the effects of colchicine on the extent of atherosclerotic plaque macrophage activity as assessed by 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Diagnosis of peripheral artery disease
3. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Use of colchicine or systemic anti-inflammatory medication (eg. tocilizumab) in the past 3 months
2. Allergy to colchicine
3. Presence of medication with drug-drug interaction
4. Acute limb ischemia requiring emergent intervention
5. Autoimmune/autoinflammatory disorders affecting blood vessels or with planned need for systemic anti-inflammatory medication
6. Recent (<14 days) systemic infection requiring hospitalization or ongoing treatment with antimicrobials
7. History of persistent anemia, thrombocytopenia, or neutropenia requiring hematology/oncology treatment or felt to pose unacceptable risk to colchicine by the principal investigator
8. Pregnant or lactating women
9. History of uncontrolled diabetes or an A1C >10% prior to the baseline visit
10. History of CrCl < 30 mL/minute or eGFR < 30mL/minute or end-stage renal disease ESRD on dialysis
11. History of liver disease or chronically-elevated (>3 months) ALT/AST > 3.0 x ULN
12. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Molecular imaging markers of inflammation | Imaging (Week 4)
  Extent of atherosclerotic plaque macrophage activity as assessed by FDG PET/CT

SECONDARY OUTCOMES:
Circulating markers of inflammation | Imaging (Week 4)
  Expression of plasma IL6 and hsCRP levels
Patient-reported walking impairment | Imaging (Week 4)
  Walking impairment as reported by Walking Impairment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No